CLINICAL TRIAL: NCT00337480
Title: A Network to Control Risk Factors After Acute Coronary Syndrome
Brief Title: Study of the Efficiency of Education About Cardiovascular Risk Factors in Patients After an Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Resicard (Other)
Responsible Party: Principal Investigator, Pr Ariel Cohen, professor, Resicard
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Resicard Prevention
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; cardiovascular risk factors; smoking habits; obesity; sedentary lifestyle; overweight; education; follow up after hospitalization
MeSH Terms: conditions — Acute Coronary Syndrome; Smoking; Obesity; Sedentary Behavior; Overweight | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional (No Intervention): This arm is the conventional way of taking care of patients after an acute coronary syndrome
- structured (Active Comparator): This arm is an active way to monitor and educate patients after their acute coronary syndrome, with the intervention of health members in a House of Education
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — education of acute coronary syndrome patients, mostly about nicotinic weaning, weight loss and physical activity
  Other Names: House of Education; Structured network; health members
  Arms: structured

SUMMARY:
The purpose of this study is to determine whether the follow up of patients with acute coronary syndrome and modifiable cardiovascular risk factors is efficient based on outpatients visits in a House of Education, underlining the importance of nicotinic weaning, weight loss and physical activity practice.

DETAILED DESCRIPTION:
1. Objectives

   1. The main purpose of this study is to evaluate the efficiency of "Resicard Prevention", which is a structured health network within a House of Education located outside of the hospital and based on outpatients' visits.
   2. Another purpose is to facilitate and optimize physicians and all health members communication around the acute coronary syndrome patients.
2. Method

   * After randomization, patients are directed to one of the two following groups: the conventional network group or the structured network group. Six and twelve months after their hospitalization, a blood test will be performed and their weight, blood pressure, waist measurement and cardiac frequency will be recorded in order to monitor patients' cardiovascular risk factors.In any case, patients receive optimal care with the participation of different health members (such as nurses, doctors, dietician...).

     a-The conventional network group
   * Patients are taken care of, according to good medical practice by their usual general practitioner and cardiologist. The frequency of consultations is set up according to symptoms. The follow up of patients is optimized as they are taken care of by a multidisciplinary health team.

     b-The structured network group
   * Patients in this group will have to consult their general practitioner and cardiologist within the first month after their hospitalization. Two forms summarizing their hospitalization facts and the objectives of the risk factors correction will be electronically sent to their general practitioner, to their cardiologist and to the House of Education. Patients have appointments at the House of Education where a multidisciplinary team (with a nurse, a dietician,...) welcomes them. They set up a schedule according to patients' needs:
   * consultation for nicotinic weaning
   * some dietary advice in order to lose weight
   * some specific advice on diabetes and/or hypercholesteremia
   * information about high blood pressure
   * some advice to pursue a regular physical activity After each appointment at the House of Education, a form summarizing the risk factors will be provided electronically to patients' general practitioner and cardiologist.
3. Conclusion -This evaluation protocol should demonstrate the efficiency of a health network based on the correction of modifiable cardiovascular risk factors within a House of Education in secondary prevention after an acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* hospitalization for acute coronary syndrome (ST segment elevation myocardial infarction, non-ST segment elevation myocardial infarction, unstable angina)
* cardiovascular risk factors during hospitalization (active and current smoking, sedentary lifestyle, obesity, overweight)
* autonomy
* agreement to visit the House of Education
* signature of a assent

Exclusion Criteria:

* lack of understanding or phrasing
* refusal to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
nicotinic weaning | 1year
weight loss at least 5% | 1 year
waist reduction at least 4% | 1 year
physical activity at least 30 minute per day (3h per week) | 1 year

SECONDARY OUTCOMES:
correction of nicotinic addiction, overweigh and lack of physical activity all together | 1 year
correction of each risk factor of primary outcome, individually | 1 year
correction of the other risk factors | 1 year
  arterial hypertension inferior to 140/90 Hgmm; low density lipoprotein cholesterol inferior to 1g/l
diabetes mellitus with HbA1C inferior to 7% | 1 year
quality of life with mental and physical scores (SF-12) | 1 year
patient's level of knowledge of the disease: number of correct answers to 19 questions | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Cohen, Pr, Principal Investigator — Hopital St Antoine
Locations (6):
- France (6):
  - Clinique la Roseraie, Aubervilliers
  - Hopital Lariboisiere, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Bichat, Paris
  - Hopital Tenon, Paris

REFERENCES:
- [Derived] Cohen A, Assyag P, Boyer-Chatenet L, Cohen-Solal A, Perdrix C, Dalichampt M, Michel PL, Montalescot G, Ravaud P, Steg PG, Boutron I; Reseau Insuffisance Cardiaque (RESICARD) PREVENTION Investigators. An education program for risk factor management after an acute coronary syndrome: a randomized clinical trial. JAMA Intern Med. 2014 Jan;174(1):40-8. doi: 10.1001/jamainternmed.2013.11342. PMID 24126705